CLINICAL TRIAL: NCT04639206
Title: A Pragmatic Trial of HOme Based Self-management & COgnitive Training CHanges Lives (HOBSCOTCH) in Georgia
Brief Title: A Pragmatic Trial of HOBSCOTCH in Georgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ngoc Cam Escoffery, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000913; CDC-STUDY00000913 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOBSCOTCH group (Experimental): Participants in this study arm will receive the HOBSCOTCH intervention immediately.
  Interventions: Behavioral: HOBSCOTCH
- Wait-listed control (No Intervention): Participants in this study arm will be wait-listed for 6 months and will then receive the HOBSCOTCH intervention.

INTERVENTIONS:
Behavioral: HOBSCOTCH — HOBSCOTCH (Home Based Self-management and Cognitive Training Changes lives) is a home-based self-management program to treat cognitive symptoms and improve quality of life while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. The HOBSCOTCH intervention consists of 8 weekly sessions conducted in-person, over the telephone, or via video-conferencing. A smart phone application will be used to collect data on seizure frequency, medication adherence, and patient engagement.
  Arms: HOBSCOTCH group

SUMMARY:
This study is being done to answer the question: Will a home-based self-management program, HOBSCOTCH, be effective in improving quality of life and perceived difficulties in cognitive abilities by teaching problem-solving strategies? The research team is also looking at a new mobile application that was developed to go with the program, and looking at extra booster sessions to improve long-term outcomes.

In order to learn about the effectiveness of the program, half of the people in this study will be randomly assigned to be in the intervention immediately. The other half will be randomly assigned to a 6-month waitlist period before getting the intervention. All participants will receive the program at some point during the study.

DETAILED DESCRIPTION:
Epilepsy affects 3.4 million people in the U.S. who suffer from many problems including seizures and medication side effects, and depression and memory problems. Epilepsy self-management programs have been proven to improve the lives of people with epilepsy (PWE). For over 10 years, the Managing Epilepsy Well (MEW) Network has developed and researched several epilepsy self-management programs with promising results. One such program is HOBSCOTCH (HOme-Based Self-management and COgnitive Training CHanges lives), which addresses memory problems and has shown improved thought processes, or cognition, in randomized control trials.

HOBSCOTCH has been tested and re-tested in the New England region with promising results in improving quality of life and cognitive functioning, or improved thought processes. To make the program more widely available, HOBSCOTCH will be offered in the state of Georgia, where the population is different compared to the New England region.

This study plans to enroll a total of 150 adults with epilepsy to participate in the program in two cycles of roughly 50-75 people. Of the 50-75 participants to enroll in the program, 25-37 participants will be assigned to the intervention group, and the other 25-37 participants will be assigned to the waitlist group. Participants will take part in the program that will last eight sessions. A trained and certified HOBSCOTCH memory coach will deliver one-on-one sessions with participants on a weekly basis and each session will last between 45-60 minutes. The first session and the last session will be done in-person or through video chat. All participants will be given standard testing at baseline, 3, 6, 9, and 12 months. The testing will help in understanding if the program helps improve memory problems and if the HOBSCOTCH program should continue to be offered to people with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy (self-reported by participant), with controlled or uncontrolled seizures
* Subjective memory complaints
* No changes in antiepileptic and antidepressant medication regimen for 1 month, however brief discontinuation of antiepileptic medicine for inpatient video electroencephalogram (EEG) evaluation is acceptable
* Literate
* Telephone access
* Internet access

Exclusion Criteria:

* Participants self-reporting a dementing illness or a dementing illness appearing in their medical record.
* Severe mental disability or estimated intelligence quotient (IQ) less than 70 per clinical judgement
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* No diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life in Epilepsy (QOLIE-31) Score | Baseline, Months 3, 6, 9, 12
  Efficacy of the HOBSCOTCH intervention will be assessed with the QOLIE-31 instrument. The QOLIE includes 31 questions about health and daily activities. Responses are given on a range of scales. Responses are coded to 0 to 100 point scales where higher scores indicate better quality of life. The final score is the average of scores for the individual items. Final scores can be converted to a T-score with a mean of 50 and standard deviation of 10, where higher T-scores indicate better quality of life.
Change in Neuro Quality of Life (Neuro-QOL) Item Bank v2.0 - Cognitive Function Score | Baseline, Months 3, 6, 9, 12
  Efficacy of the HOBSCOTCH intervention will be assessed with the Neuro-QOL instrument.The Neuro-QOL - Cognitive Function questionnaire includes 28 items asking about how much difficulty they are experiencing and how often they have had trouble with certain tasks during the past 7 days. Responses are given on a scale from 1 to 5 where 1 = cannot do/very often and 5 = none/never. Total scores range from 28 to 140 and higher scores indicate improved cognitive function.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire - 9 Depression (PHQ-9) Score | Baseline, Months 3, 6, 9, 12
  The PHQ-9 is a 9-item instrument assessing symptoms of depression in the prior two weeks. Responses are given on a 4-point scale where 0 = not at all and 3 = nearly everyday. Total scores range from 0 to 27 where higher scores indicate greater feelings of depression.
Change in Adult Epilepsy Self-Management Measurement Instrument (AESMMI-65) Score | Baseline, Months 3, 6, 9, 12
  The AESMMI-65 is a 65-item instrument assessing 11 domains of self-management of epilepsy. Responses are given on a 5-point scale where 1 = none of the time and 5 = all of the time. Certain items are reverse scored and total scores range from 65 to 325, where higher scores indicate better practice of self-management behaviors.
Seizure Frequency | Baseline to Month 12
  Seizure frequency will be assessed by a self-reported daily log completed either with the mobile application or paper log.
Change in Medication Adherence Rating Scale (MARS) Score | Baseline, Months 3, 6, 9, 12
  The MARS is a 10-item instrument asking about behaviors and attitudes related to medications. Responses of "yes" are scored as 0 and responses of "no" are scored as 1. Total scores range from 0 to 10 where higher scores indicate greater medication adherence.
Change in Health Confidence Score (HCS) | Baseline, Months 3, 6, 9, 12
  Participants are asked four questions assessing their confidence in their own health care. Responses are scored on a 4-point scale where 0 = disagree and 3 = strongly agree. Total scores range from 0 to 12 where higher scores indicate greater confidence regarding health care.
Change in Health Care Utilization | Baseline, Months 3, 6, 9, 12
  Participants will be asked to report their utilization of health care in the prior 6 months.
Change in Well-being | Baseline to Month12
  Daily well-being will be assessed via the mobile app for a paper log. Participants will rate their well-being as Great, Good, Average, Poor, or Very Poor.

CONTACTS AND LOCATIONS:
Overall Officials: Cam Escoffery, PhD, MPH, Principal Investigator — Emory University; Katie Bullinger, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Brain Health Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04639206/ICF_000.pdf